CLINICAL TRIAL: NCT03112174
Title: Phase 3 Study of Ibrutinib in Combination With Venetoclax in Subjects With Mantle Cell Lymphoma
Brief Title: Study of Ibrutinib Combined With Venetoclax in Subjects With Mantle Cell Lymphoma (MCL)
Acronym: SYMPATICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCYC-1143-CA; 2017-000129-12 (EudraCT Number)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Mantle-Cell Lymphoma
Keywords: PCYC; MCL; Non-Hodgkin's Lymphoma; NHL; ibrutinib; venetoclax; Pharmacyclics
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-in (Experimental): Participants with a low or high risk of TLS enroll into the open-label Safety Run-in Period to receive concurrent ibrutinib at 560 mg once daily and venetoclax starting at 20 mg, and gradually ramp up to a target dose of 400 mg once daily over a 5-week period.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Randomization Phase: Ibrutinb + Venetoclax (Experimental): Participants randomized to ibrutinib and venetoclax for approximately 104 weeks, followed by ibrutinib monotherapy until disease progression (PD), unacceptable toxicity or withdrawal of consent. Venetoclax is discontinued after 104 weeks of treatment, regardless of response assessment.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Randomization Phase: Ibrutinib + Placebo (Placebo Comparator): Participants randomized to ibrutinib and placebo for approximately 104 weeks, followed by ibrutinib monotherapy until PD, unacceptable toxicity or withdrawal of consent. Placebo is discontinued after 104 weeks of treatment, regardless of response assessment.
  Interventions: Drug: Ibrutinib; Drug: Placebo Oral tablet to match Venetoclax
- Treatment-naive Open-label Arm (Experimental): Participants are treated with ibrutinib 560 mg and venetoclax 400 mg, administered using the 5-week ramp-up schedule.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Administered orally once daily
Drug: Venetoclax — Administered orally once daily
  Arms: Randomization Phase: Ibrutinb + Venetoclax; Safety Run-in; Treatment-naive Open-label Arm
Drug: Placebo Oral tablet to match Venetoclax — Administered orally once daily
  Arms: Randomization Phase: Ibrutinib + Placebo

SUMMARY:
This Phase 3 multinational, randomized, double-blind study is designed to compare the efficacy and safety of the combination of ibrutinib and venetoclax vs. ibrutinib and placebo in subjects with MCL.

ELIGIBILITY:
Relapsed/Refractory Arm

Inclusion Criteria:

* Pathologically confirmed MCL (in tumor tissue), with documentation of either overexpression of cyclin D1 in association with other relevant markers (eg, CD19, CD20, PAX5, CD5) or evidence of t(11;14) as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR).
* At least 1 measurable site of disease on cross-sectional imaging (CT).
* At least 1, but no more than 5, prior treatment regimens for MCL.
* Failure to achieve at least partial response (PR) with, or documented disease progression after, the most recent treatment regimen.
* Subjects must have adequate fresh or paraffin embedded tissue.
* Adequate hematologic, hepatic and renal function.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of <= 2.

Exclusion Criteria:

* History or current evidence of central nervous system lymphoma.
* Concurrent enrollment in another therapeutic investigational study or prior therapy with ibrutinib or other BTK inhibitors.
* Prior treatment with venetoclax or other BCL2 inhibitors.
* Anticancer therapy including chemotherapy, radiotherapy, small molecule and investigational agents <= 21 days prior to receiving the first dose of study drug.
* Treatment with any of the following within 7 days prior to the first dose of study drug: moderate to strong cytochrome P450 3A (CYP3A) inhibitors or strong CYP3A inducers.

Treatment Naïve Arm

Inclusion Criteria:

* Pathologically confirmed treatment-naive MCL (tumor tissue), with documentation of either overexpression of cyclin D1 in association with other relevant markers (eg, CD19, CD20, PAX5, CD5) or evidence of t(11;14), as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR).
* Men and women ≥18 years of age with a TP53 mutation.
* At least 1 measurable site of disease by CT.
* Must have adequate fresh or paraffin-embedded tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 to <= 2.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Blastoid variant of MCL
* History or current evidence of CNS lymphoma.
* Concurrent enrollment in another therapeutic investigational study or prior therapy including ibrutinib or other BTK inhibitors.
* Prior treatment with venetoclax or other BCL2 inhibitors.
* Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study drug.
* Clinically significant infection requiring IV systemic treatment that was completed <=14 days before the first dose of study drug.
* Any uncontrolled active systemic infection.
* Known bleeding disorders (eg, von Willebrand's disease or hemophilia).
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* History of HIV or active HCV or HBV.
* Major surgery within 4 weeks of the first dose of study drug.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the participant's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Unable to swallow capsules or tablets, or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Treatment with any of the following within 7 days prior to the first dose of study drug: Moderate or strong cytochrome P450 3A (CYP3A) inhibitors or moderate or strong CYP3A inducers.
* Known allergy to xanthine oxidase inhibitors and/or rasburicase for subjects with known risk factors (as defined by high tumor burden and/or diminished renal function, as detailed in "Study Design" section above) for TLS.
* Chronic liver disease with hepatic impairment Child-Pugh class B or C.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Known hypersensitivity to the active ingredient or other components of one or more study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (120):
- United States (14):
  - The University of Arizona Cancer Centre-North Campus, Tucson, Arizona
  - City of Hope, Duarte, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - Orlando Health Inc., Orlando, Florida
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - University of Tennessee medical Center, Knoxville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (7):
  - The Canberra Hospital, Canberra, Australian Capital Territory
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Icon Cancer Care, Auchenflower, Queensland
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer, Melbourne, Victoria
  - St.Vincent's Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (4):
  - ZiekenhuisNetwerk Antwerpen (ZNA) Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Institut Jules Bordet, Brussels
  - CHU UCL Namur asbl- Mont Godinne, Yvoir
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer-Vancouver Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Czechia (6):
  - FN Brno, Interni hematologicka a onkologicka klinika, Brno
  - Fakultni Nemocnice (FN) Hradec Kravlove, a.s. IV. Interni hematologicka klinika, Hradec Králové
  - FN Olomouc, Olomouc
  - FN Ostrava, Ostrava-Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, l. interni klinika-klinika hematologie, Prague
- France (8):
  - CHU CAEN-Hôpital de la Côte de Nacre, Caen, Calvados
  - Institut Bergonié, Bordeaux
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Institut Paoli Calmettes, Service Hematologie, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Tours, Tours
- Germany (10):
  - Kliniken Ostalb Stauferklinikum Schwab. Gmund, Mutlangen, Baden-Wuttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wuttemberg
  - Klinikum der Universitaet Muenchen Campus Grosshadern, Munich, Bavaria
  - Universitatsklinikum Koln, Kerpen, Koln
  - Universitaetsmedizin der Johannes Gutenberg, Langenbeckstrasse 1, Langen, Mainz
  - Gemeinschaftpraxis Haematologie und Onkologie, Dresden, Saxony
  - Vivantes Klinikum Am Urban, Berlin
  - Charite- Universitatsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Essen, Klinik fur Hamatologie, Essen
  - Universitatsklinikum des Saarlandes, Klinik fur Innere Medizin I, Homburg/Saar
- Greece (7):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - 251 Air Force General Hospital, Athens
  - General Hospital of Athens Laiko, Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
- Hungary (7):
  - Orszagos Onkologiai Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, II. Belgyogyaszat-Hematologia, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Haematologiai es Haemoszatazeologiai Osztaly, Szombathely
- Italy (11):
  - Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria, Alessandria/Piemonte
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Bergamo/Lombardia
  - Azienda Ospedaliera Universitaria di Bologna Policlinico Saint Orsola Malpighi, Bologna, Bologna/Emilia-Romagna
  - ASST degli Spedali Civili di Brescia, Brescia, Brescia/Lombardia
  - Azienda Ospedaliera S. Croce e Carle Cuneo, Cuneo, Cuneo/Piemonte
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Forli-Cesena/Emilia-Rom
  - IRCCS Ospedale S. Raffaele di Milano, Milan, Milano/Lombardia
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Milano/Lombardia
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia/Lombardia
  - Azienda Ospedaliero Universitaria Molinette San Giovanni Battista di Torino, Torino, Torino/Piemonte
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine, Udine/Friuli-Venezia Giulia
- Netherlands (5):
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Gasthuis, Hoofddorp
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam
  - Franciscus Vlietland, Schiedam
- Poland (6):
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela w Bydgoszcz, Bydgoszcz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Oddzial Hematologiczny, Chorzów
  - Malopolskie Centrum Medyczne s c, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. Kopernika w Lodzi, Lodz
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu, PZOZ, Wroclaw
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (7):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - ICO l'Hospitalet- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cabuenes, Gijón, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
- Turkey (Türkiye) (4):
  - Ondokuz Mayiz universitesi Tip Fakultesi, Kurupelit, Samsun
  - Gazi Universitesi Tip Fakultesi, Besevler, Ankara
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Namik Kemal Universitesi Saglik Uyg. ve.Ars. Hastanesi, Tekirdağ
- Ukraine (6):
  - Communal Nonprofit enterprise Cherkasy Regional Oncology Dispensary ofCherkasy Oblast Council,Regional Treatment and Diagnostic Hematological Center, Cherkasy
  - Communal Non-profit Enterprise Regional Center of Oncology, Department of Hematology, Kharkiv
  - National Inst. of Cancer, Scientific and Research Dept of Chemotherapy of Hemoblastosis and Adjuvant Treatment Methods, Dept of Oncohematology with Sector of Adjuvant treatment methods, Kyiv
  - SI national Scientific Center of Radiation Medicine of NAMS of Ukraine, Dep. of Radiation Oncohematology and Stem Cell Transplantation Unit, Kyiv
  - Andrii Novak Transcarpathian Regional Clinical Hospital, Department of Hematology, Uzhhorod
  - Communal Institution O.F. Herbachevskyi Regional Clinical Hospital of Zhytomyr Regional Council Dept of Hematology with beds of Intensive Therapy, Zhytomyr
- United Kingdom (7):
  - Barts Health NHS Trust, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - The Churchill Hospital, Oxford, Oxfordshire
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - St James University Hospital, Leeds, West Yorkshire
  - University College London Hospitals NHS Foundation Trust, London

REFERENCES:
- [Derived] Wang M, Jurczak W, Trneny M, Belada D, Wrobel T, Ghosh N, Keating MM, van Meerten T, Alvarez RF, von Keudell G, Thieblemont C, Peyrade F, Andre M, Hoffmann M, Szafer-Glusman E, Lin J, Dean JP, Neuenburg JK, Tam CS. Ibrutinib plus venetoclax in relapsed or refractory mantle cell lymphoma (SYMPATICO): a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2025 Feb;26(2):200-213. doi: 10.1016/S1470-2045(24)00682-X. PMID 39914418
- [Derived] Wang M, Ramchandren R, Chen R, Karlin L, Chong G, Jurczak W, Wu KL, Bishton M, Collins GP, Eliadis P, Peyrade F, Lee Y, Eckert K, Neuenburg JK, Tam CS. Concurrent ibrutinib plus venetoclax in relapsed/refractory mantle cell lymphoma: the safety run-in of the phase 3 SYMPATICO study. J Hematol Oncol. 2021 Oct 30;14(1):179. doi: 10.1186/s13045-021-01188-x. PMID 34717692

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Run-in: Increased TLS Risk at Baseline: Participants with an increased risk of tumor lysis syndrome (TLS) enrolled into the open-label Safety Run-in Period received concurrent ibrutinib at 560 mg once daily and venetoclax starting at 20 mg, and gradually ramped up to a target dose of 400 mg once daily over a 5-week period.
- Safety Run-in: Low TLS Risk at Baseline: Participants with an low risk of TLS enrolled into the open-label Safety Run-in Period received concurrent ibrutinib at 560 mg once daily and venetoclax starting at 20 mg, and gradually ramped up to a target dose of 400 mg once daily over a 5-week period.
- Randomization Phase: Ibrutinb + Venetoclax: Participants were randomized to ibrutinib 560 mg and venetoclax (starting at 20 mg, and gradually ramped up to a target dose of 400 mg) once daily over a 5-week period for approximately 104 weeks, followed by ibrutinib monotherapy until disease progression (PD), unacceptable toxicity or withdrawal of consent. Venetoclax was discontinued after 104 weeks of treatment, regardless of response assessment.
- Randomization Phase: Ibrutinib + Placebo: Participants were randomized to ibrutinib 560 mg and placebo for approximately 104 weeks, followed by ibrutinib monotherapy until PD, unacceptable toxicity or withdrawal of consent. Placebo was discontinued after 104 weeks of treatment, regardless of response assessment.
- Treatment-naive Open-label Arm: Participants were treated with ibrutinib 560 mg and venetoclax (starting at 20 mg, and gradually ramped up to a target dose of 400 mg).
Period: Overall Study
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Started | 15 | 6 | 134 | 133 (1 participant in this arm did not receive any dose of study drug.) | 78
On Study Treatment at Study Closure | 0 | 2 | 31 | 21 | 26
Off Treatment and On Study Follow Up at Study Closure | 2 | 0 | 22 | 25 | 25
Completed (Completed=Participants followed for progression (if not progressed before treatment discontinuation), subsequent anticancer therapy, and survival status until study closure. Not Completed=Already off study at study closure.) | 2 | 2 | 53 | 46 | 51
Not Completed | 13 | 4 | 81 | 87 | 27
Not completed — Withdrawal by Subject | 3 | 0 | 11 | 9 | 7
Not completed — Lost to Follow-up | 1 | 1 | 2 | 3 | 2
Not completed — Death | 8 | 3 | 67 | 73 | 18
Not completed — Other, Not Specified | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomization Phase: Ibrutinb + Venetoclax: Participants were randomized to ibrutinib 560 mg and venetoclax (starting at 20 mg, and gradually ramped up to a target dose of 400 mg) for approximately 104 weeks, followed by ibrutinib monotherapy until disease progression (PD), unacceptable toxicity or withdrawal of consent. Venetoclax was discontinued after 104 weeks of treatment, regardless of response assessment.
- Total: Total of all reporting groups
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm | Total
Number analyzed (Participants) | 15 | 6 | 134 | 133 | 78 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 41 | 47 | 13 | 108
  >=65 years | 13 | 1 | 93 | 86 | 65 | 258
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 31 | 25 | 25 | 89
  Male | 9 | 4 | 103 | 108 | 53 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 8 | 7 | 1 | 17
  Not Hispanic or Latino | 11 | 5 | 112 | 110 | 72 | 310
  Unknown or Not Reported | 3 | 1 | 14 | 16 | 5 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 3 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 3
  White | 12 | 6 | 116 | 115 | 68 | 317
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 15 | 14 | 3 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Lysis Syndrome (TLS) Events (Safety Run-in)
Description: TLS events are defined as follows:
  * Clinical TLS: any event that meets Howard criteria (N Engl J Med 2011;364:1844-1854) with the following exceptions:
    * For the purpose of TLS assessment during the Safety Run-in Period, only those increases in serum creatinine > 1.0 mg/dL from pre-treatment baseline will be considered clinical TLS.
    * In participants with renal dysfunction at baseline (CrCl < 60 mL/min), clinical TLS is defined as the presence of laboratory TLS plus either seizures, cardiac dysrhythmia, or death.
  * Laboratory TLS: any event that meets Howard criteria (N Engl J Med 2011;364:1844-1854) for laboratory TLS, that does not resolve within 72 hours despite protocol required management.
Time Frame: After at least 3 months of treatment, with an overall median treatment duration of 20.0 months
Population: All treated safety run-in participants
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
Participants | 1 | 0

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) (Safety Run-in)
Description: DLT: any Grade (Gr) 3 or higher non-TLS adverse event (AE) at least possibly related to study drug occurring during the DLT assessment period with the following clarifications:
  Non-Hematologic DLTs: Gr ≥3 nausea, vomiting or diarrhea uncontrolled despite maximum medical supportive care and persisting >5 days; Gr 3 fatigue persisting >7 days; Gr 3 infection is not a DLT, however an infection with lifethreatening consequences or requiring urgent intervention (Gr 4) was considered a DLT; Treatment delay of any study drug >7 days for toxicity.
  Hematologic DLTs: Gr 3 neutropenia is not a DLT, however, Gr 4 neutropenia (ANC <500/mm^3) lasting for > 7 days is a DLT; Gr 3 or 4 neutropenia complicated by fever ≥38.5°C or infection; Gr 4 thrombocytopenia (<25,000/mm^3) that persists for > 7 days; Gr 3 or 4 thrombocytopenia associated with Gr 2 or greater bleeding; Gr 3 anemia is not a DLT, however, Gr 4 anemia is a DLT; Treatment delay of any study drug >7 days for hematologic toxicity.
Time Frame: After at least 3 months of treatment, with an overall median treatment duration of 20.0 months
Population: All treated safety run-in participants
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
Participants
  Any TEAE/Any Grade | 3 | 0
  Any TEAE/ Grade 3+4 | 3 | 0
  Any TEAE/Grade 5 | 0 | 0
  Atrial fibrillation/Any Grade | 1 | 0
  Atrial fibrillation/Grade 3+4 | 1 | 0
  Atrial fibrillation/Grade 5 | 0 | 0
  Infection/Any Grade | 1 | 0
  Infection/Grade 3+4 | 1 | 0
  Infection/Grade 5 | 0 | 0
  Neutropenia/Any Grade | 1 | 0
  Neutropenia/Grade 3+4 | 1 | 0
  Neutropenia/Grade 5 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) (Safety Run-in)
Description: AE: any untoward medical occurrence in a participant that does not necessarily have a causal relationship with treatment. The investigator assesses the relationship of each event to the use of study. Serious adverse event (SAE): an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs): any event that began or worsened in severity on or after the first dose of study drug. Event severity is graded as mild (1), moderate (2), severe (3), life threatening (4), death (5).
Time Frame: From first dose of study drug until the end of treatment + 30 days, with an overall median treatment duration of 20.0 months
Population: All treated safety run-in participants
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
Participants
  Any TEAE | 15 | 6
  Any TEAE, Grade 3 | 15 | 5
  Any Venetoclax (V) Related TEAE | 14 | 6
  Any V Related TEAE Grade >=3 | 13 | 4
  Any Ibrutinib (I) Related TEAE | 13 | 5
  Any I Related TEAE Grade >=3 | 12 | 4
  Any TEAE Leading to Discontinuation of Study Drug (I or V) | 6 | 2
  Any TEAE Leading to Discontinuation of Study Drug (I only) | 1 | 0
  Any TEAE Leading to Discontinuation of Study Drug (V only) | 1 | 0
  Any TEAE Leading to Discontinuation of Study Drug (Both I and V) | 4 | 2
  Any TEAE Leading to Dose Reduction of Study Drug (I or V) | 7 | 4
  Any TEAE Leading to Dose Reduction of Study Drug (I Only) | 1 | 3
  Any TEAE Leading to Dose Reduction of Study Drug (V Only) | 3 | 0
  Any TEAE Leading to Dose Reduction of Study Drug (Both I and V) | 3 | 1
  Any TEAE Leading to Dose Hold of Study Drug (I or V) | 14 | 4
  Any TEAE Leading to Dose Hold of Study Drug (I Only) | 1 | 1
  Any TEAE Leading to Dose Hold of Study Drug (V Only) | 0 | 0
  Any TEAE Leading to Dose Hold of Study Drug (Both I and V) | 13 | 3
  Any TESAE | 14 | 3
  Any TESAE, Grade >=3 | 14 | 2
  Any TESAE, V Related | 9 | 1
  Any TESAE, I Related | 10 | 1
  Any TESAE, V or I Related | 10 | 1
  Fatal TEAE | 1 | 0
  Major Hemorrhage | 2 | 0
  Major Hemorrhage, Grade >=3 | 2 | 0
  Major Hemorrhage, TESAE | 2 | 0

4. Primary Outcome: Progression-free Survival (PFS) (Randomization Phase)
Description: PFS is defined as the time from the date of randomization to the date of disease progression using the Revised Response Criteria for Malignant Lymphoma (Cheson 2014), or death from any cause, whichever occurs first.
Time Frame: For an overall median time on study of 61.34 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Randomization Phase: Ibrutinb + Venetoclax: Participants were randomized to ibrutinib 560 mg and venetoclax (starting at 20 mg, and gradually ramped up to a target dose of 400 mg) for approximately 104 weeks, followed by ibrutinib monotherapy until PD, unacceptable toxicity or withdrawal of consent. Venetoclax was discontinued after 104 weeks of treatment, regardless of response assessment.
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 134 | 133
months | 31.9 [22.8 to 54.5] | 22.1 [16.5 to 29.5]
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.0024, Log Rank — P value is from stratified log-rank test; Hazard Ratio (HR) = 0.629, 95% CI 2-sided [0.465 to 0.850]

5. Primary Outcome: Complete Response (CR) Rate (Treatment-Naive Arm)
Description: CR rate is defined as the percentage of participants with a CR according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2014).
Time Frame: For an overall median time on study of 40.51 months
Population: All Enrolled Treatment-Naïve Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment-naive Open-label Arm
Number analyzed (Participants) | 78
percentage of participants | 69.2 [57.8 to 79.2]

6. Secondary Outcome: Overall Survival (OS) (Safety Run-in)
Description: OS is defined as the time from the date of the first dose of study treatment to death from any cause.
Time Frame: For an overall median time on study of 74.78 months
Population: All Enrolled Safety Run-in participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
months | 52.3 [14.1 to NA] — Not estimable due to small number of events. | NA [1.5 to NA] — Not estimable due to small number of events.

7. Secondary Outcome: Progression-free Survival (PFS) (Safety Run-in)
Description: PFS is defined as the time from the date of the first dose of study treatment to the date of disease progression using the Revised Response Criteria for Malignant Lymphoma (Cheson 2014), or death from any cause, whichever occurs first.
Time Frame: For an overall median time on study of 74.78 months
Population: All Enrolled Safety Run-in participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
months | 46.9 [13.0 to NA] — Not estimable due to the small number of events. | 35.0 [1.2 to NA] — Not estimable due to the small number of events.

8. Secondary Outcome: Duration of Response (DOR) (Safety Run-in)
Description: DOR is defined for participants who achieve an overall response as the time from the first occurrence of response (CR or PR according to the Revised Response Criteria for Malignant Lymphoma [Cheson 2014]) to disease progression or death, whichever occurs first.
Time Frame: For an overall median time on study of 74.78 months
Population: All Enrolled Safety Run-in Subjects Achieving Response (Partial Response or Better)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 12 | 5
months | 44.1 [12.5 to NA] — Not estimable due to the small number of events. | NA [26.5 to NA] — Not estimable due to the small number of events.

9. Secondary Outcome: Overall Response Rate (ORR) (Safety Run-in)
Description: ORR is defined as the percentage of participants with CR or PR per investigator assessment according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2014).
Time Frame: For an overall median time on study of 74.78 months
Population: All enrolled Safety Run-in participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline
Number analyzed (Participants) | 15 | 6
percentage of participants | 80.0 [51.9 to 95.7] | 83.3 [35.9 to 99.6]

10. Secondary Outcome: Percentage of Participants With a Complete Response (CR) (Randomization Phase)
Description: Complete response rate (CR) based on the best overall response per investigator assessment according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2014).
Time Frame: For an overall median time on study of 61.34 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 134 | 133
percentage of participants | 53.7 [44.9 to 62.4] | 32.3 [24.5 to 41.0]
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — Estimate and p-value for rate ratio are based on Cochran-Mantel-Haenszel (CMH) test adjusted for two randomization stratification factors: number of prior lines of therapy (1-2 vs >=3) and TLS category (low risk vs increased risk) at randomization; Rate Ratio = 1.658, 95% CI 2-sided [1.240 to 2.218] — For rate ratio, numerator is Ibrutinib + Venetoclax arm and denominator is Ibrutinib + Placebo arm

11. Secondary Outcome: Overall Response Rate (ORR) (Randomization Phase and Treatment-Naive Arm)
Description: as for outcome 9
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase) and 40.51 months (Treatment-Naïve arm)
Population: All randomized participants and all treatment-naive open-label arm participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Number analyzed (Participants) | 134 | 133 | 78
percentage of participants | 82.1 [74.5 to 88.2] | 74.4 [66.2 to 81.6] | 94.9 [87.4 to 98.6]
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.1279, Cochran-Mantel-Haenszel — Estimate and p-value for rate ratio are based on CMH test adjusted for two randomization stratification factors: number of prior lines of therapy (1-2 vs >=3) and TLS category (low risk vs increased risk) at randomization; Rate Ratio = 1.101, 95% CI 2-sided [0.973 to 1.247] — For rate ratio, numerator is Ibrutinib + Venetoclax arm and denominator is Ibrutinib + Placebo arm

12. Secondary Outcome: MRD-negative Remission Rate in Participants Who Achieve CR Per Investigator Assessment (Randomization Phase and Treatment-Naive Arm)
Description: MRD-negative remission rate is defined as the percentage of participants with undetectable MRD at documented CR in participants who were MRD positive at screening as assessed by flow cytometry in bone marrow and/or peripheral blood, with requirement of confirmation of MRD negativity in the subsequent peripheral blood 12 weeks later.
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase) and 40.51 months (Treatment-Naïve arm)
Population: All enrolled treatment-naïve participants achieving CR who were evaluable for MRD (those who had positive MRD status at screening). Participants with a given post-screening sample.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Number analyzed (Participants) | 31 | 8 | 34
percentage of participants
  Bone marrow aspirate: number analyzed (Participants) | 26 | 7 | 22
  Bone marrow aspirate | 61.5 [40.6 to 79.8] | 28.6 [3.7 to 71.0] | 59.1 [36.4 to 79.3]
  Peripheral blood | 77.4 [58.9 to 90.4] | 12.5 [0.3 to 52.7] | 76.5 [58.8 to 89.3]
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Bone marrow aspirate; Test type: Superiority; p = 0.2028, Fisher Exact
Statistical Analysis 2: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Peripheral blood; Test type: Superiority; p = 0.0014, Fisher Exact

13. Secondary Outcome: Overall Survival (OS) (Randomization Phase and Treatment-Naive Arm)
Description: OS is defined as the time from the date of randomization (Randomization Phase) or the first dose of study treatment (Treatment-Naïve arm) to death from any cause.
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase) and 40.51 months (Treatment-Naïve arm)
Population: All randomized and all enrolled treatment-naïve participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Number analyzed (Participants) | 134 | 133 | 78
months | 44.9 [31.9 to NA] — Not estimable due to the small number of events. | 38.6 [25.2 to 52.6] | NA [44.2 to NA] — Not estimable due to the small number of events.
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.2669, Log Rank — P value is from stratified log-rank test; Hazard Ratio (HR) = 0.832, 95% CI 2-sided [0.602 to 1.151] — Hazard ratio is estimated using stratified Cox regression model with treatment as the only covariate

14. Secondary Outcome: Duration of Response (DOR) (Randomization Phase and Treatment-Naive Arm)
Description: DOR is defined as the time frame for participants who achieve an overall response as the time from the first occurrence of response (CR or PR according to the Revised Response Criteria for Malignant Lymphoma [Cheson 2014]) to disease progression or death, whichever occurs first.
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase) and 40.51 months (Treatment-Naïve arm)
Population: All randomized participants and all enrolled treatment-naïve participants achieving response (partial response or better)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment-naive Open-label Arm: Participants were treated withibrutinib 560 mg and venetoclax (starting at 20 mg, and gradually ramped up to a target dose of 400 mg).
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Number analyzed (Participants) | 110 | 99 | 74
months | 42.1 [28.7 to NA] — Not estimable due to the small number of events. | 27.6 [19.4 to 39.5] | 37.1 [30.3 to NA] — Not estimable due to the small number of events.

15. Secondary Outcome: Time to Next Treatment (TTNT) (Randomization Phase and Treatment-Naive Arm)
Description: TTNT is defined as the duration from the date of randomization (Randomization Phase) or date of first dose of study treatment (Treatment-Naive Arm) to the start date of any anti-lymphoma treatment subsequent to study treatment. Post-treatment stem cell transplantation, chimeric antigen receptor (CAR) T-cell therapy, or other cellular therapies were not considered subsequent anti-cancer treatments for participants responding to the study treatment (CR or PR).
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase) and 40.51 months (Treatment-Naïve arm)
Population: All randomized and all enrolled treatment-naïve participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
Number analyzed (Participants) | 134 | 133 | 78
months | NA [48.0 to NA] — Not estimable due to the small number of events | 35.4 [24.7 to 49.8] | NA [NA to NA] — Not estimable due to the small number of events
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.0013, Log Rank — P value is from stratified log-rank test; Hazard Ratio (HR) = 0.541, 95% CI 2-sided [0.369 to 0.792] — Hazard ratio is estimated using stratified Cox regression model with treatment as the only covariate

16. Secondary Outcome: Number of Participants With TEAEs (Randomization Phase)
Description: as for outcome 3
Time Frame: From first dose of study drug until the end of treatment + 30 days, with an overall median treatment duration of 19.5 months
Population: All randomized and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 134 | 132
Participants
  Any TEAE | 134 | 131
  Any TEAE, Grade 3 | 113 | 100
  Any Venetoclax (V) Related TEAE | 112 | 104
  Any V Related TEAE Grade >=3 | 75 | 46
  Any Ibrutinib (I) Related TEAE | 121 | 114
  Any I Related TEAE Grade >=3 | 83 | 58
  Any TEAE Leading to Discontinuation of Study Drug (I or V) | 43 | 48
  Any TEAE Leading to Discontinuation of Study Drug (I only) | 15 | 11
  Any TEAE Leading to Discontinuation of Study Drug (V only) | 2 | 7
  Any TEAE Leading to Discontinuation of Study Drug (Both I and V) | 26 | 30
  Any TEAE Leading to Dose Reduction of Study Drug (I or V) | 50 | 29
  Any TEAE Leading to Dose Reduction of Study Drug (I Only) | 19 | 14
  Any TEAE Leading to Dose Reduction of Study Drug (V Only) | 13 | 7
  Any TEAE Leading to Dose Reduction of Study Drug (Both I and V) | 18 | 8
  Any TEAE Leading to Dose Hold of Study Drug (I or V) | 106 | 99
  Any TEAE Leading to Dose Hold of Study Drug (I Only) | 18 | 18
  Any TEAE Leading to Dose Hold of Study Drug (V Only) | 6 | 4
  Any TEAE Leading to Dose Hold of Study Drug (Both I and V) | 82 | 77
  Any TESAE | 88 | 80
  Any TESAE, Grade >=3 | 76 | 73
  Any TESAE, V Related | 31 | 25
  Any TESAE, I Related | 47 | 37
  Any TESAE, V or I Related | 49 | 37
  Fatal TEAE | 22 | 18
  Major Hemorrhage | 13 | 8
  Major Hemorrhage, Grade >=3 | 10 | 7
  Major Hemorrhage, TESAE | 12 | 6

17. Secondary Outcome: Number of Participants With TLS TEAEs (Randomization Phase)
Description: Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs): any event that began or worsened in severity on or after the first dose of study drug (SD). Event severity is graded as mild (1), moderate (2), severe (3), life threatening (4), death (5).
Time Frame: From first dose of study drug until the end of treatment + 7 days, with an overall median treatment duration 19.5 months
Population: All randomized and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 134 | 132
Participants
  Any Grade | 7 | 3
  Grades 3 and 4 | 6 | 3

18. Secondary Outcome: Steady-State Pharmacokinetics (PK) of Ibrutinib: Maximum Observed Plasma Concentration (Cmax) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: Week 6, Day 1: Predose, at Dose, 1 hour (± 15 minutes [min]), 2 hours (± 15 min), 4 hours (± 30 min), 6 hours (± 30 min), 8 hours (± 1 hour), 24 hours post-dose
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 106 | 108
ng/mL | 195 (179) | 287 (230)

19. Secondary Outcome: Steady-State PK of Ibrutinib: Time to Cmax (Tmax) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 106 | 108
hours | 2.00 [0.00 to 8.00] | 2.00 [0.750 to 6.00]

20. Secondary Outcome: Steady-State PK of Ibrutinib: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 102 | 106
ng·h/mL | 1090 (870) | 1440 (1060)

21. Secondary Outcome: Steady-State PK of Ibrutinib: Terminal Elimination Half-Life (t1/2,Term) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 65 | 73
hours | 6.29 (1.92) | 6.66 (2.15)

22. Secondary Outcome: Steady-State PK of Ibrutinib: Time of Last Measurable Concentration (Tlast) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 102 | 106
hours | 24.0 [7.0 to 24.0] | 24.0 [24.0 to 24.0]

23. Secondary Outcome: Steady-State PK of Ibrutinib: Area Under the Concentration-Time Curve From 0-24 Hours (AUC0-24) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 102 | 106
ng·h/mL | 1090 (870) | 1440 (1060)

24. Secondary Outcome: Steady-State PK of Ibrutinib: Terminal Elimination Rate Constant (λz) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 65 | 73
1/hour | 0.123 (0.0556) | 0.114 (0.0332)

25. Secondary Outcome: Steady-State PK of Ibrutinib: Apparent Total Clearance at Steady State (CLss/F) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 102 | 106
L/hour | 1020 (1130) | 709 (651)

26. Secondary Outcome: Steady-State PK of Venetoclax: Cmax (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants receiving venetoclax with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax
Number analyzed (Participants) | 102
ng/mL | 3620 (1650)

27. Secondary Outcome: Steady-State PK of Venetoclax: AUC0-24 (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants receiving venetoclax with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax
Number analyzed (Participants) | 98
ng·h/mL | 65000 (32900)

28. Secondary Outcome: Steady-State PK of Venetoclax: Time to Cmax (Tmax) (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants receiving venetoclax with an evaluable PK assessment at given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax
Number analyzed (Participants) | 102
hours | 6.00 [0.00 to 8.03]

29. Secondary Outcome: Steady-State PK of Venetoclax: CLss/F (Randomization Phase)
Description: Pre-dose concentrations were applied as 24-hour concentrations in order to calculate steady-state PK parameters.
Time Frame: as for outcome 18
Population: Participants receiving venetoclax with an evaluable PK assessment at given time point.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax
Number analyzed (Participants) | 98
L/hour | 8.09 (4.82)

30. Secondary Outcome: Time to Worsening in Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale of the Health-related Quality of Life (Randomization Phase)
Description: The FACT-Lym lymphoma-specific additional concerns subscale responses to all items are rated on a 5-point scale ranging from 0 "not at all" to 4 "very much". The lymphoma subscale includes 15 items and scores range from 0 to 60, with higher scores representing better functional status and well-being. A 5-point change in the Lym subscale was selected as a conservative estimate of clinically meaningful deterioration in lymphoma symptoms.
Time Frame: For an overall median time on study of 61.34 months (Randomization Phase)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo
Number analyzed (Participants) | 134 | 133
months | 9.3 [6.5 to 12.7] | 12.5 [8.3 to 17.9]
Statistical Analysis 1: Comparison: Randomization Phase: Ibrutinb + Venetoclax vs Randomization Phase: Ibrutinib + Placebo; Test type: Superiority; p = 0.2861, Log Rank — P value is from stratified log-rank test; Hazard Ratio (HR) = 1.169, 95% CI 2-sided [0.879 to 1.554]

31. Secondary Outcome: Duration of CR (Treatment-Naive Arm)
Description: Duration of CR, defined for subjects who achieve CR according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2014) as the time from the first occurrence of CR to disease progression or death, whichever occurs first.
Time Frame: For an overall median time on study of 40.51 months
Population: All Enrolled Treatment-Naïve Subjects Achieving CR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment-naive Open-label Arm
Number analyzed (Participants) | 54
months | 37.1 [34.0 to NA] — Not estimable due to low number of events.

32. Secondary Outcome: Progression-free Survival (PFS) (Treatment-Naive Arm)
Description: as for outcome 7
Time Frame: For an overall median time on study of 40.51 months
Population: All enrolled treatment-naïve participants
Measure: Median (Full Range); unit: months
Arm/Group | Treatment-naive Open-label Arm
Number analyzed (Participants) | 78
months | 40.2 [29.4 to NA] — Not estimable due to low number of events.

ADVERSE EVENTS:
Time Frame: For an overall median duration of 69.6 months (Safety Run-in: Increased TLS Risk), 77.9 months (Safety Run-in: Low TLS Risk), 61.0 months (Randomization Phase: Ibrutinb + Venetoclax), 61.7 months (Randomization Phase: Ibrutinb + Placebo), 40.5 months (Treatment-naive Open-label Arm).
Description: All treated participants
Groups:
- Safety Run-in: Increased TLS Risk at Baseline: Participants with an increased risk of TLS enrolled into the open-label Safety Run-in Period received concurrent ibrutinib at 560 mg once daily and venetoclax starting at 20 mg, and gradually ramped up to a target dose of 400 mg once daily over a 5-week period.
Arm/Group | Safety Run-in: Increased TLS Risk at Baseline | Safety Run-in: Low TLS Risk at Baseline | Randomization Phase: Ibrutinb + Venetoclax | Randomization Phase: Ibrutinib + Placebo | Treatment-naive Open-label Arm
All-Cause Mortality (participants affected / at risk) | 8/15 | 3/6 | 70/134 | 78/132 | 20/78
Serious Adverse Events (participants affected / at risk) | 15/15 | 3/6 | 92/134 | 86/132 | 48/78
Other Adverse Events (participants affected / at risk) | 15/15 | 6/6 | 131/134 | 127/132 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-in: Increased TLS Risk at Baseline (N=15) | Safety Run-in: Low TLS Risk at Baseline (N=6) | Randomization Phase: Ibrutinb + Venetoclax (N=134) | Randomization Phase: Ibrutinib + Placebo (N=132) | Treatment-naive Open-label Arm (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 6 (7) | 2 (2) | 0 (0)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
SPONTANEOUS HAEMORRHAGE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (10) | 4 (4) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 0 (0) | 6 (7) | 3 (4) | 3 (3)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (3)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MITRAL VALVE DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 3 (5)
SEROSITIS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ANTI-NEUTROPHIL CYTOPLASMIC ANTIBODY POSITIVE VASCULITIS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GRAFT VERSUS HOST DISEASE IN GASTROINTESTINAL TRACT (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
CENTRAL NERVOUS SYSTEM INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 6 (10) | 1 (1) | 8 (11)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (7) | 2 (4) | 6 (7)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DISSEMINATED CRYPTOCOCCOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FUNGAL ABSCESS CENTRAL NERVOUS SYSTEM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MEDIASTINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (3) | 0 (0) | 17 (26) | 15 (17) | 5 (6)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA CHLAMYDIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA MORAXELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 7 (7) | 2 (3) | 1 (1)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 15 (23) | 18 (27) | 1 (1)
MANTLE CELL LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRADYKINESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 2 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (6) | 6 (6) | 0 (0)
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOSS OF PERSONAL INDEPENDENCE IN DAILY ACTIVITIES (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-in: Increased TLS Risk at Baseline (N=15) | Safety Run-in: Low TLS Risk at Baseline (N=6) | Randomization Phase: Ibrutinb + Venetoclax (N=134) | Randomization Phase: Ibrutinib + Placebo (N=132) | Treatment-naive Open-label Arm (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 4 (20) | 2 (2) | 27 (40) | 17 (32) | 17 (27)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 12 (17) | 10 (12) | 17 (25)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 12 (53) | 1 (2) | 2 (2)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (33) | 1 (2) | 46 (207) | 19 (25) | 26 (67)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 4 (5) | 22 (74) | 20 (46) | 8 (23)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 12 (14) | 12 (16) | 10 (10)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 5 (8) | 3 (3) | 7 (10)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 3 (5)
ASTIGMATISM (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 2 (2) | 0 (0) | 5 (6) | 9 (9) | 3 (5)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (5) | 2 (2)
DRY EYE (Eye disorders) | 4 (4) | 2 (3) | 18 (25) | 20 (45) | 8 (14)
EYE DISCHARGE (Eye disorders) | 1 (1) | 1 (1) | 2 (3) | 5 (5) | 2 (2)
EYE IRRITATION (Eye disorders) | 2 (5) | 1 (2) | 13 (16) | 21 (27) | 6 (6)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 6 (10) | 7 (10) | 1 (1)
HYPERMETROPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 2 (2) | 2 (6) | 18 (30) | 16 (25) | 9 (15)
MACULAR DEGENERATION (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MACULOPATHY (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 3 (3) | 1 (3) | 11 (14) | 12 (19) | 3 (4)
PHOTOPSIA (Eye disorders) | 2 (2) | 0 (0) | 5 (8) | 3 (3) | 1 (1)
VISION BLURRED (Eye disorders) | 4 (5) | 3 (10) | 25 (47) | 23 (50) | 8 (17)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (3) | 1 (1) | 20 (42) | 16 (32) | 9 (13)
VITREOUS FLOATERS (Eye disorders) | 2 (2) | 2 (3) | 5 (7) | 10 (12) | 5 (6)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (4) | 1 (1) | 14 (22) | 12 (17) | 11 (20)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (8) | 9 (11) | 7 (8)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (9) | 5 (10)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 2 (5) | 19 (23) | 23 (59) | 13 (19)
DIARRHOEA (Gastrointestinal disorders) | 10 (24) | 5 (21) | 84 (243) | 48 (89) | 37 (196)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (9) | 10 (11) | 3 (4)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 19 (28) | 11 (13) | 8 (12)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 3 (7) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECES SOFT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMORAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (6) | 3 (3) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8) | 5 (6) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 11 (15) | 5 (5) | 11 (12)
GLOSSODYNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 7 (10) | 3 (3) | 4 (4)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 2 (3) | 11 (15) | 6 (6) | 7 (13)
NAUSEA (Gastrointestinal disorders) | 5 (15) | 5 (16) | 43 (78) | 21 (36) | 24 (75)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
PEPTIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (2) | 1 (3) | 12 (16) | 11 (20) | 12 (31)
TONGUE ERYTHEMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONGUE HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
VOMITING (Gastrointestinal disorders) | 5 (9) | 1 (11) | 27 (59) | 14 (24) | 18 (35)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (3) | 0 (0) | 26 (38) | 18 (24) | 6 (12)
CATHETER SITE BRUISE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 6 (7) | 4 (5) | 1 (1)
CHILLS (General disorders) | 2 (2) | 2 (2) | 8 (8) | 4 (4) | 4 (6)
EXTRAVASATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 5 (12) | 4 (12) | 39 (66) | 36 (77) | 30 (78)
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 10 (11) | 5 (6) | 4 (4)
INJECTION SITE BRUISING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 3 (4) | 16 (20) | 21 (28) | 14 (15)
PAIN (General disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 6 (6)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 1 (1) | 11 (19) | 9 (11) | 3 (9)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 28 (51) | 28 (56) | 16 (20)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (2) | 1 (7) | 2 (10) | 2 (3) | 0 (0)
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (7) | 1 (1) | 6 (8)
PORTAL FIBROSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 7 (10) | 9 (15) | 4 (5)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 1 (3) | 0 (0) | 8 (10) | 11 (15) | 3 (3)
COVID-19 (Infections and infestations) | 2 (4) | 1 (1) | 16 (20) | 16 (22) | 19 (22)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (13) | 2 (3) | 5 (5) | 2 (2)
DEMODICIDOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPIDIDYMITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (2)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 8 (10) | 5 (6)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 7 (12) | 2 (2) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 5 (8) | 1 (1) | 2 (4)
NASAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 8 (11) | 8 (9) | 4 (4)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 8 (10) | 7 (9) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (2) | 5 (6) | 7 (12) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 7 (7) | 7 (9) | 2 (3)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 6 (11) | 7 (18) | 2 (3)
RHINITIS (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 9 (10) | 2 (2)
SINUSITIS (Infections and infestations) | 1 (2) | 0 (0) | 11 (14) | 6 (8) | 4 (8)
SKIN CANDIDA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINEA CRURIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (2) | 23 (42) | 14 (16) | 9 (13)
URINARY TRACT INFECTION (Infections and infestations) | 4 (14) | 1 (4) | 14 (22) | 10 (12) | 7 (21)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 8 (8) | 3 (3) | 6 (7)
FALL (Injury, poisoning and procedural complications) | 4 (6) | 1 (1) | 11 (11) | 7 (7) | 6 (9)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (5)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 5 (6) | 2 (2) | 2 (2)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 5 (7) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 1 (3) | 4 (4) | 3 (5) | 4 (9)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 1 (3) | 5 (5) | 2 (2) | 5 (11)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (3) | 4 (7) | 1 (1) | 1 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (2) | 2 (6) | 3 (4) | 2 (4) | 3 (19)
BLOOD CREATININE INCREASED (Investigations) | 3 (6) | 2 (3) | 7 (8) | 13 (27) | 7 (9)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 7 (9) | 2 (2) | 2 (2)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 2 (2) | 5 (12) | 10 (32)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 0 (0) | 3 (3) | 5 (11) | 6 (10)
TROPONIN T INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (4) | 0 (0) | 15 (17) | 7 (7) | 6 (7)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (4) | 2 (2) | 3 (3)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 24 (33) | 15 (18) | 8 (9)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 8 (8)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 9 (12)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (3) | 9 (12) | 11 (15) | 5 (5)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (11) | 2 (2) | 21 (31) | 8 (13) | 16 (24)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 (5) | 4 (6) | 14 (23) | 4 (13) | 16 (21)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (3) | 4 (5) | 1 (4)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 4 (5) | 4 (6) | 4 (7)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 4 (5) | 3 (3) | 4 (4)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (8) | 22 (29) | 23 (47) | 12 (26)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 12 (18) | 15 (20) | 14 (26)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 4 (6) | 4 (10) | 3 (3)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 12 (16) | 32 (56) | 6 (10)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (7) | 1 (5) | 1 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (13) | 13 (18) | 17 (34) | 16 (34)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 11 (18) | 12 (18) | 8 (14)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 7 (10) | 5 (5) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (21) | 16 (22) | 20 (35) | 17 (23)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 4 (4)
DYSKINESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 3 (4) | 15 (19) | 22 (43) | 15 (21)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (4) | 8 (10) | 6 (9) | 7 (19)
MEMORY IMPAIRMENT (Nervous system disorders) | 3 (3) | 1 (1) | 1 (3) | 4 (10) | 2 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (3) | 5 (9) | 14 (23) | 9 (19)
PARESIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 7 (13) | 6 (8)
PRESYNCOPE (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (5) | 2 (2)
SENSORY DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 6 (7) | 3 (4) | 1 (1)
TREMOR (Nervous system disorders) | 2 (3) | 0 (0) | 2 (4) | 1 (1) | 2 (2)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 1 (1) | 5 (6) | 6 (7) | 4 (5)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 2 (2) | 12 (12) | 13 (14) | 9 (10)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (4) | 0 (0)
BLADDER HYPERTROPHY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (7) | 4 (5) | 6 (8)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (5) | 5 (7) | 11 (13)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (5) | 2 (3) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (3) | 4 (4) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 28 (46) | 35 (55) | 13 (17)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (3) | 17 (24) | 15 (24) | 14 (23)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (7) | 9 (14) | 14 (23) | 6 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 7 (8) | 6 (6) | 4 (5)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 14 (15) | 15 (21) | 3 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 5 (8) | 6 (7) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (7) | 0 (0)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 3 (3) | 1 (1)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 6 (7) | 5 (5) | 4 (4)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 7 (8) | 3 (3) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 9 (10) | 5 (6) | 2 (2)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (13) | 7 (9) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (8) | 5 (10) | 7 (11)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 15 (18) | 15 (26) | 11 (13)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (7) | 2 (3) | 2 (2)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 8 (9) | 5 (6) | 5 (5)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (6) | 18 (33) | 12 (14) | 13 (19)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (7) | 1 (1) | 3 (4)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (2) | 5 (12)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (4) | 1 (5) | 20 (32) | 23 (28) | 15 (23)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 7 (7) | 4 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03112174/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03112174/SAP_001.pdf